CLINICAL TRIAL: NCT06493812
Title: Comparison of Clinical Value in the Use of the Fascia Lata and Temporal Muscle Fascia in the Reconstruction of the Dura in the Sellar Region
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klinički Bolnički Centar Zagreb (Other)
Responsible Party: Principal Investigator, Marcel Marjanovic Kavanagh, Principal investigator, Klinički Bolnički Centar Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/013 AG
Record Dates: First submitted 2024-06-30; First posted 2024-07-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Skull Defect; Transplant Complication; Quality of Life
Keywords: CSF; fascia lata; temporal fascia; quality of life; tissue transplantation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia lata (Active Comparator): Participants in this group will undergo skull base reconstruction using fascia lata harvested from the thigh. The surgical team will perform endoscopic endonasal surgery to treat sellar region pathology and utilize fascia lata to repair the skull base defect. The procedure involves the extraction of the graft from the left thigh, followed by standard reconstruction techniques to ensure optimal healing and function of the skull base. Postoperative pain and other outcomes will be closely monitored and recorded using standardized measures.
  Interventions: Procedure: Fascia lata
- Temporal fascia (Active Comparator): Participants in this group will undergo skull base reconstruction using temporal muscle fascia harvested from the temporal region of the head. The surgical team will perform endoscopic endonasal surgery to treat sellar region pathology and utilize temporal fascia to repair the skull base defect. The procedure involves the extraction of the graft from the left temporal region, followed by standard reconstruction techniques to ensure optimal healing and function of the skull base. Postoperative pain and other outcomes will be closely monitored and recorded using standardized measures.
  Interventions: Procedure: Temporal fascia

INTERVENTIONS:
Procedure: Fascia lata — This intervention involves the harvesting of fascia lata from the thigh and its use in reconstructing the skull base defect following endoscopic endonasal surgery for sellar region pathology. The graft is extracted from the left thigh, and standard reconstruction techniques are employed to ensure optimal healing and functionality of the skull base. Postoperative monitoring includes assessments of donor site pain, incidence of complications, and overall recovery using standardized measures.
  Arms: Fascia lata
Procedure: Temporal fascia — This intervention involves the harvesting of temporal muscle fascia from the temporal region of the head and its use in reconstructing the skull base defect following endoscopic endonasal surgery for sellar region pathology. The graft is extracted from the left temporal region, and standard reconstruction techniques are employed to ensure optimal healing and functionality of the skull base. Postoperative monitoring includes assessments of donor site pain, incidence of complications, and overall recovery using standardized measures.
  Arms: Temporal fascia

SUMMARY:
Study Title: Assessing the Clinical Significance of Using Fascia Lata versus Temporalis Muscle Fascia for Skull Base Reconstruction in Sellar Region

Objective: The primary objective of this study is to investigate and compare the effectiveness and safety of using fascia lata and temporal muscle fascia in the reconstruction of the skull base in the sellar region. Specifically, the study aims to determine and compare the level of donor site pain between the two groups using Visual Analogue Scales (VAS). The study also aims to identify the optimal method and materials for skull base reconstruction that result in the lowest frequency of complications, thereby reducing perioperative morbidity and enabling earlier rehabilitation of patients.

Subjects and Methods:

Study Design: Prospective randomized controlled trial. Population: The study will enroll 68 patients who have undergone endoscopic endonasal surgery for sellar region pathology. Patients will be divided into two groups: one group will receive skull base reconstruction using fascia lata, and the other group will receive reconstruction using temporal fascia.

Interventions: In the fascia lata group, grafts will be harvested from the thigh, while in the temporal fascia group, grafts will be harvested from the temporal muscle area.

Measurements:

Primary Outcome: Donor site pain measured using Visual Analogue Scales (VAS) at various postoperative intervals (preoperative, and on the 1st, 2nd, and 3rd postoperative days, as well as 1 month and 3 months post-surgery).

Secondary Outcomes: Incidence of postoperative complications such as meningitis, cerebrospinal fluid (CSF) leak, donor site infection, and other surgical complications.

Expected Contribution: This research is expected to provide valuable insights into the comparative effectiveness and safety of using fascia lata versus temporal muscle fascia for skull base reconstruction. The findings could influence clinical decisions regarding the choice of graft material, potentially leading to reduced perioperative morbidity, faster patient rehabilitation, and improved overall outcomes for patients undergoing skull base surgeries.

DETAILED DESCRIPTION:
Study Title: Assessing the Clinical Significance of Using Fascia Lata versus Temporalis Muscle Fascia for Skull Base Reconstruction in Sellar Region

Study Objective: The primary objective of this prospective randomized controlled study is to evaluate and compare the effectiveness and safety of using fascia lata and temporal muscle fascia for skull base reconstruction in the sellar region following endoscopic endonasal surgery. The study aims to determine the level of donor site pain using Visual Analogue Scales (VAS) and to identify the optimal reconstruction method with the lowest complication rates.

Background: Tumors in the sellar region, such as pituitary adenomas, craniopharyngiomas, meningiomas, and chordomas, present significant surgical challenges due to their location. Advances in endoscopic techniques have improved surgical outcomes for these tumors, but complications, particularly cerebrospinal fluid (CSF) leaks, remain common. Reconstruction of skull base defects is critical to prevent CSF leaks and associated infections. Autologous grafts, including fascia lata and temporal muscle fascia, are commonly used for this purpose. This study seeks to compare these two graft materials in terms of effectiveness, safety, and patient quality of life post-surgery.

Study Design:

Type: Prospective randomized controlled trial. Enrollment: 68 adult patients.

Randomization: Participants will be randomly assigned to one of two groups:

Group 1: Skull base reconstruction using fascia lata. Group 2: Skull base reconstruction using temporal muscle fascia. Blinding: Single-blind (patients will not know which type of fascia is used for their reconstruction).

Duration: The study will commence in August 2023 and is expected to last for 2-3 years.

Inclusion Criteria:

Adult patients (18 years and older) undergoing endoscopic endonasal surgery for sellar region tumors.

Patients requiring reconstruction of the sellar floor to prevent postoperative CSF leaks.

Exclusion Criteria:

Pathology at the donor site (trauma, previous surgery). Absence of intraoperative CSF leak. Use of alternative reconstruction materials. Prior radiation therapy to the operative or donor site.

Interventions:

Group 1 (Fascia Lata): Grafts harvested from the thigh. Group 2 (Temporal Fascia): Grafts harvested from the temporal muscle area. All surgeries will be performed by a standardized surgical team comprising a neurosurgeon and an otolaryngologist. The techniques for incision, hemostasis, and reconstruction will be consistent across all procedures.

Outcome Measures:

Primary Outcome:

Donor site pain assessed using Visual Analogue Scales (VAS) at the following time points: preoperative, postoperative days 1, 2, and 3, and at 1 and 3 months post-surgery.

Secondary Outcomes:

Incidence of postoperative complications such as meningitis, CSF leak, donor site infection, wound dehiscence, seroma, facial nerve palsy, hypoesthesia of the donor site skin, and diabetes insipidus (temporary or permanent).

Quality of life measured using the EQ-5D-5L questionnaire before surgery and at 1 and 3 months postoperatively.

Duration of surgical procedures. Length of hospital stay.

Statistical Analysis:

Power Analysis: A sample size of 34 participants per group is required to achieve 80% power to detect a 30% difference in the incidence of mild versus moderate/severe pain (VAS > 3.5), with a significance level of α = 0.05. Power analysis was conducted using MedCalc® Statistical Software version 22.003.

Data Analysis: Normality of data distribution will be tested using histograms and the Kolmogorov-Smirnov test. Continuous variables will be presented as mean (95% confidence interval) or median (interquartile range), depending on distribution. Categorical variables will be presented as absolute frequencies and percentages. Differences in continuous variables between groups will be analyzed using one-way ANOVA with post-hoc tests for parametric data or Kruskal-Wallis test with Dunn's post-hoc test for non-parametric data. Differences in categorical variables will be analyzed using Fisher-Freeman-Halton test for independent samples or McNemar's test for paired samples. A significance level of p < 0.05 will be considered statistically significant. Data analysis will be performed using IBM SPSS Statistics version 29.0.1.

Ethical Considerations:

The study has been approved by the Ethics Committee of KBC Zagreb. Informed consent will be obtained from all participants prior to their inclusion in the study.

Participant privacy will be protected by anonymizing personal data and using unique coded identifiers. Access to anonymized data will be strictly controlled, and any de-anonymization will occur only under the supervision of the Ethics Committee.

Funding: The study is funded through clinical research funds dedicated to scientific investigations at KBC Zagreb.

Expected Contributions: The study aims to provide empirical evidence on the comparative effectiveness and safety of fascia lata versus temporal muscle fascia for skull base reconstruction. Results will guide clinical decision-making, potentially reducing perioperative morbidity, enhancing patient recovery, and improving quality of life post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. **Age**: Adult patients (18 years and older).
2. **Surgical Requirement**: Patients undergoing endoscopic endonasal surgery for sellar region tumors requiring reconstruction of the sellar floor to prevent postoperative cerebrospinal fluid (CSF) leaks.
3. **Consent**: Patients who provide informed consent to participate in the study.

Exclusion Criteria:

* 1. **Donor Site Pathology**: Presence of pathology at the donor site, including trauma or previous surgical interventions.

  2. **Absence of Intraoperative CSF Leak**: Patients without an intraoperative CSF leak requiring reconstruction.

  3. **Alternative Reconstruction Methods**: Use of reconstruction materials other than fascia lata or temporal fascia.

  4. **Prior Radiation Therapy**: Patients who have received prior radiation therapy to the operative or donor site.

  5. **Medical Contraindications**: Patients with medical conditions that contraindicate the surgical procedure or participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2033-08-01 (Estimated); Study Completion 2033-12-01 (Estimated)

PRIMARY OUTCOMES:
Donor Site Pain | Preoperative, Postoperative Days 1, 2, and 3, and at 1 month and 3 months post-surgery.
  The primary outcome measure is the level of donor site pain, assessed using Visual Analogue Scales (VAS).
  Visual Analog Scale (VAS) for Pain
  Minimum Value: 0 (No pain) Maximum Value: 10 (Worst pain imaginable)
  Outcome Interpretation Higher scores indicate worse outcomes (more intense pain).
  The VAS is a simple and widely used tool to help patients quantify their pain level. Patients mark their pain level on a 10 cm line that ranges from "no pain" to "worst pain imaginable."

SECONDARY OUTCOMES:
Incidence of Postoperative Complications | Up to 3 months post-surgery.
  The frequency of complications following the surgical procedures, including:
  * Meningitis
  * Postoperative cerebrospinal fluid (CSF) leak
  * Donor site wound dehiscence
  * Donor site infection
  * Seroma formation at the donor site
  * Facial nerve palsy
  * Hypoesthesia of the donor site skin
  * Diabetes insipidus (temporary or permanent)
Quality of life - EQ 5D | Preoperative, 1 month post-surgery, and 3 months post-surgery.
  Assessment of the patients' quality of life using the EQ-5D-5L questionnaire.
  * **Minimum Value**: The EQ-5D-5L generates a descriptive profile and a single index value. For the descriptive profile, each of the 5 dimensions has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The single index value ranges from -0.281 (theoretical minimum, country-specific) to 1 (perfect health).
  * **Outcome Interpretation**: Higher scores on the descriptive profile indicate worse health states. For the single index value, higher scores indicate better health outcomes.
  The EQ-5D-5L is used to assess the general health status of a patient across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels of severity, and the responses can be combined into a single index value representing overall health status.

CONTACTS AND LOCATIONS:
Locations (1):
- KBC Zagreb, Zagreb, Croatia